CLINICAL TRIAL: NCT00214149
Title: A UW Phase II Trial of Multi-catheter HDR Brachytherapy Following Lumpectomy for Early Stage Breast Breast Cancer
Brief Title: Multi-catheter High Dose Rate (HDR) Breast Brachytherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lost funding
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RO04102; 2004-0268 (Other: Institutional Review Board)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): breast brachytherapy to a dose of 34 Gy
  Interventions: Radiation: brachytherapy

INTERVENTIONS:
Radiation: brachytherapy — breast brachytherapy to 34 Gy

SUMMARY:
Breast conservation therapy (BCT) is now widely accepted as a treatment option for most women with Stage I and II invasive breast cancer and most patients with ductal carcinoma in situ (DCIS). Despite superior cosmetic outcome, BCT is more complex and requires a protracted treatment regimen comprised of 6 weeks of daily external beam radiation therapy to the whole breast. The purpose of this study is to determine if an acceptable outcome can be achieved with radiation delivered only to the region of the tumor bed. If this is true, partial breast irradiation may lend itself to much shorter treatment times (one week) and the toxicities to adjacent normal structures (heart, lung, chest wall) will be greatly reduced.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer or DCIS, tumor stage of Tis, T1, T2 if lesion is < 3 cm, N0 or N1 if 1-3 + nodes with no extracapsular extension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Patel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] McHaffie DR, Patel RR, Adkison JB, Das RK, Geye HM, Cannon GM. Outcomes after accelerated partial breast irradiation in patients with ASTRO consensus statement cautionary features. Int J Radiat Oncol Biol Phys. 2011 Sep 1;81(1):46-51. doi: 10.1016/j.ijrobp.2010.05.011. Epub 2010 Aug 21. PMID 20732760

RESULTS

PARTICIPANT FLOW:
Groups:
- Breast Brachytherapy to 34 Gy: breast brachytherapy to a dose of 34 Gy
  brachytherapy: breast brachytherapy to 34 Gy
Period: Overall Study
Arm/Group | Breast Brachytherapy to 34 Gy
Started | 127
Completed | 0 (No data are available; study was terminated and PI has left the institution.)
Not Completed | 127

BASELINE CHARACTERISTICS:
Arm/Group | Breast Brachytherapy to 34 Gy
Number analyzed (Participants) | 127
Age, Customized [Number; unit: years]
  Age 30-39 | 2
  Age 40-49 | 29
  Age 50-59 | 35
  Age 60-69 | 45
  Age 70-79 | 14
  Age 80-89 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 123
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 124
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 127

OUTCOME MEASURES:

1. Primary Outcome: To Determine if Brachytherapy Will Produce Non-inferior Local Regional Control at 5 Years Post Treatment When Compared to Historical Results of Conventional XRT
Time Frame: 5 years
Population: No data are available as the study was terminated and PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed. Sincere efforts were made to obtain the data for reporting, however, no data are available.
Arm/Group | Breast Brachytherapy to 34 Gy
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine if Brachytherapy Will Produce Non-inferior Toxicity to XRT at 3 Years
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Breast Brachytherapy to 34 Gy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study was terminated early, adverse events data were collected on paper that presumably are with the PI.
Description: No data are available as the study was terminated and PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed. Sincere efforts were made to obtain the data for reporting, however, no data are available.
Arm/Group | Breast Brachytherapy to 34 Gy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
We were able to find a published paper that may represent some of the results of this study (linked in the references section of the protocol). The number of participants does not match our records as our records for this study are incomplete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-12-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT00214149/Prot_SAP_000.pdf